CLINICAL TRIAL: NCT04397744
Title: Unidas Por Vida y Salud: Increasing Breast and Cervical Cancer Screening in El Paso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Maria E Fernandez, Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-12-0677
Record Dates: First submitted 2020-05-17; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer; Cervical Cancer
Keywords: Mammogram; Pap test
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unidas por Vida y Salud prevention program (Experimental): Unidas por Vida y Salud (United for Life and Health) prevention program
  Interventions: Behavioral: Unidas por Vida y Salud prevention program
- No intervention control (No Intervention): The control arm will not receive the Unidas por Vida y Salud (United for Life and Health) prevention program during the study analysis period (though, the control arm will receive the intervention after study has been completed).

INTERVENTIONS:
Behavioral: Unidas por Vida y Salud prevention program — The Unidas por Vida y Salud (United for Life and Health) prevention program is led by the El Paso Cancer and Chronic Disease Consortium (CCDC), the only Breast and Cervical Cancer Services (BCCS) provider in El Paso. This prevention program will use a well-integrated network of community organizations and health service providers to connect medically underserved women to services. To reach the most underserved women and increase preventive cancer screening and timely follow-up, diagnosis, and treatment, the multi-method approach uses evidence-based strategies, including face-to-face educational sessions led by promotoras (community health workers), client reminders, and provision of community-based navigation services to affordable and free screening services. The program also includes clinic-based navigation for those requiring diagnostics or treatment delivered by trained nurses and case workers.
  Arms: Unidas por Vida y Salud prevention program

SUMMARY:
The purpose of this study is to develop, implement and evaluate a comprehensive breast and cervical cancer screening program designed to increase uptake of breast and cervical cancer screening among rarely and never-screened low-income women in El Paso County and to increase repeat screening among those currently overdue.

ELIGIBILITY:
Inclusion Criteria:

* overdue for a repeat mammogram
* overdue for repeat cervical screening

Exclusion Criteria:

-

Ages: 21 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 660 (Actual)
Dates: Start 2015-01-16 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Number of participants who uptake clinical breast exam (CBE) | 6 months
Number of participants who uptake mammography | 6 months
Number of participants who uptake pap test | 6 months
Number of participants who repeat mammography | 6 months
Number of participants who repeat pap test | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Fernandez, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Savas LS, Atkinson JS, Figueroa-Solis E, Valdes A, Morales P, Castle PE, Fernandez ME. A lay health worker intervention to improve breast and cervical cancer screening among Latinas in El Paso, Texas: A randomized control trial. Prev Med. 2021 Apr;145:106446. doi: 10.1016/j.ypmed.2021.106446. Epub 2021 Feb 4. PMID 33548363